CLINICAL TRIAL: NCT06725524
Title: A Phase 1, Open-Label, Multi-center Study Evaluating the Safety and Tolerability of of JMT601 in Participants With Relapsed or Refractory CD20-positive B-cell Non-Hodgkin Lymphoma
Brief Title: A Study of JMT601 in Participants With Relapsed or Refractory CD20-positive B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT601-001
Record Dates: First submitted 2023-07-19; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JMT601 (Experimental): Subjects will receive JMT601 once a week. The first 4-week period is for DLT observation.
  Dose escalation part will be carried out according to 3+3 dose-escalation design with up to 6 dose(0.3 mg/kg, 1 mg/kg, 3 mg/kg, 6 mg/kg, 12 mg/kg and 20 mg/kg) escalation cohorts.
  Dose expansion part will continue at the determined RP2D. Dose expansion part consists of two cohorts:
  Cohort A: Subjects with CD20-positive diffuse large B-cell lymphoma, prior at least two lines of therapy.
  Cohort B: Subjects with CD20-positive follicular lymphoma, prior at least two lines of therapy.
  Interventions: Biological: JMT601

INTERVENTIONS:
Biological: JMT601 — intravenous infusion on day 1 once a week

SUMMARY:
This is a Phase 1, open-label, multi-center study to evaluate the safety of JMT601 in the treatment of relapsed or refractory CD20-positive B-cell non-Hodgkin lymphoma and to determine the recommended dose for Phase 2 studies (RP2D). Study consists of 2 parts. The first part is a dose-escalation part using a 3+3 design with up to 6 dose(0.3 mg/kg, 1 mg/kg, 3 mg/kg, 6 mg/kg, 12 mg/kg and 20 mg/kg) escalation cohorts at increasing levels. The second part is a dose-expansion part at R2PD dose to assess preliminary efficacy of JMT601.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants diagnosed with CD20-positive B-cell non-Hodgkin lymphoma confirmed by histopathology and/or cell biology who have previously received 2 or more lines of therapy
* Eastern Cooperative Oncology Group (ECOG) physical state score: 0-2
* Participants must have at least one evaluable or measurable lesion according to Lugano 2014 criteria.
* Expected survival of at least 3 months;
* Suitable organ and hematopoietic function:

  1. The absolute count of neutrophil (ANC) ≥1.0×109/L;
  2. Platelets ≥75×10^9/L (if bone marrow invasion doesn't exist)/≥50.0×10^9/L (if bone marrow invasion exists);
  3. Hemoglobin ≥90 g/L;
  4. Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min;
  5. Total bilirubin ≤1.5×ULN, alanine aminotransferase ≤2.5×ULN, aspartate aminotransferase ≤2.5×ULN; Subjects with liver lesion: TBIL≤3×ULN, ALT≤5×ULN, AST≤5×ULN;
  6. International Standardized ratio and activated partial thromboplastin time ≤1.5 × ULN;

Key Exclusion Criteria:

* Confirmed central nervous system (CNS) lymphoma.
* Subjects who have received allogeneic hematopoietic stem cell transplantation (HSCT) or other organ transplantation
* Those who have previously received targeted CD47 or signal regulatory protein α (SIRRP α) therapy.
* Previous or current hemolytic anemia, Evans syndrome, arteritis;
* Subjects with previous or current other malignant tumors;
* Previous or current history of active autoimmune diseases;
* Subjects who had undergone major surgery within 4 weeks prior to initial dosing or expected to have major surgery during the study period;
* HIV infection, active syphilis, hepatitis B surface antigen (HBsAg) positive and HBV-DNA higher than the lower limit or 1000 copies /ml(500 IU/ml), HCV antibody positive and HCV-RNA higher than the lower limit or 1000 copies /ml

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) and maximum tolerated dose(MTD) | DLTs and MTD: Up to 28 days after the first dose
Incidence of treatment-emergent adverse events (TEAEs) | TEAEs: Up to 90 days after last dose

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 12 months
  Defined as the proportion of participants with complete response or partial response measured by Lugano 2014
Duration of response (DOR) | Up to 12 months
  Defined as the time from complete response or partial response to progression disease or death
Progression free survival (PFS) | Up to 12 months
  Defined as the time from initiation of treatment to progression disease or death
Overall survival (OS) | Up to 12 months
  Defined as the time from initiation of treatment to death of any cause
Aera under the curve from 0 to the last measurable concentration(AUClast) | Up to 12 months
  Aera under the curve from 0 to the last measurable concentration
Aera under the curve from 0 to the infinite time(AUC0-∞) | Up to 12 months
  Aera under the curve from 0 to the infinite time
Time to maximum concentration(Tmax) | Up to 12 months
  time to maximum concentration
Terminal phase half-life(T1/2) | Up to 12 months
  terminal phase half-life
Clearance(CL) | Up to 12 months
  clearance
Volume(Vd) | Up to 12 months
  volume
Maximum concentration( Cmax) | Up to 12 months
  maximum concentration
Minimum concentration(Cmin) | Up to 12 months
  minimum concentration
Accumulation ratio(AR) | Up to 12 months
  accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Principal Investigator — Ruijin Hospital Clinical, Shanghai Jiao Tong University, School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No